CLINICAL TRIAL: NCT07034391
Title: A Phase II Single-Arm Study Evaluating the Efficacy of PD-1 Inhibitor Combined With Denosumab and Chemotherapy in Locally Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer Patients With Driver Gene-Negative Status
Brief Title: A Study Evaluating the Efficacy of PD-1 Inhibitor Combined With Denosumab and Chemotherapy in Locally Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer Patients With Driver Gene-Negative Status
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Xiujuan Qu, Chief Physician, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-NSCLC-LUDX-3001
Record Dates: First submitted 2025-05-18; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- denosumab combined chemotherapy plus anti-PD-1/PD-L1 inhibitor (Experimental)
  Interventions: Drug: denosumab combined anti-PD-1 inhibitor with chemotherapy

INTERVENTIONS:
Drug: denosumab combined anti-PD-1 inhibitor with chemotherapy — 120mg of denosumab，d1 in a 28-days cycle；200mg of anti-PD-1 inhibitor, d1 in a 21-days cycle；500mg/m2 of pemetrexed, d1 in a 21-days cycle; AUC4-5 of carboplatin, d1 in a 21-days cycle, for 4-6 cycle

SUMMARY:
This is an interventional study to explore the efficacy and safety of denosumab combined chemotherapy and anti-PD-1/PD-L1 inhibitor in locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC)
* Documented negative for EGFR/ALK/ROS1/BRAFV600E/RET/METex14 mutations by validated genomic testing, with no prior targeted therapy and no history of other malignancies
* No previous systemic therapy for advanced/metastatic disease
* At least one measurable lesion per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* No use of parathyroid hormone/derivatives, calcitonin, osteoprotegerin, mithramycin, or potassium supplements within the past 6 months
* Adequate organ and marrow function

Exclusion Criteria:

* Histologically or cytologically confirmed combined small cell and non-small cell lung cancer (mixed histology)
* Any previous systemic anticancer treatment for NSCLC, including chemotherapy, biologics, immunotherapy, or investigational agents
* Prior use of denosumab or any bone-modifying agents (e.g., bisphosphonates)
* Uncontrolled hypocalcemia or hypophosphatemia
* History or current evidence of osteonecrosis of the jaw (ONJ) or osteomyelitis of the jaw

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | 6 months
  6-month progression-free rate

SECONDARY OUTCOMES:
progression-free survival（PFS） | 24 months
overall survival (OS) | 24 months
objective response rate (ORR) | 6 months
disease control rate (DCR) | 6 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Qu chief physician, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China